CLINICAL TRIAL: NCT01203800
Title: Evaluation of Blood Brain Barrier Permeability in Chronic Stroke
Status: Completed | Type: Observational
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Principal Investigator, Mordechai Lorberboym Prof, PI, Wolfson Medical Center
Other Study IDs: 0056-09-WOMC
Record Dates: First submitted 2010-09-15; First posted 2010-09-16 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-02

CONDITIONS: A Positive or a Negative Brain SPECT

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In this study the investigators intend to explore the long term significance of BBB disruption on the clinical course and the rate of significant recurrent ischemic events in patients with a chronic stroke.

DETAILED DESCRIPTION:
Evaluation of Blood Brain Barrier Permeability in Chronic Stroke

Mordechai Lorberboym, M.D.1, Yair Lampl, M.D.2, Ronit Gilad, M.D.2.

From the Department of Nuclear Medicine1 and the department of Neurology2 of the Edith Wolfson Medical Center, Sackler Faculty of Medicine, Tel Aviv University, Tel Aviv, Israel.

Introduction

The blood brain barrier (BBB) is a highly selective barrier of brain microvascular endothelial cells that shields the brain from toxic substances in the blood, supplies brain tissues with nutrients, and filters harmful compounds from the brain back to the bloodstream (1). Transport across the BBB is strictly limited through both physical (tight junctions) and metabolic barriers (enzymes, diverse transport systems). BBB breakdown or alterations in transport systems play an important role in the pathogenesis of many CNS diseases (HIV-1 encephalitis, Alzheimer's disease, ischemia, tumors, multiple sclerosis, and Parkinson's disease).

Cerebral ischemia leads to disruption of blood flow, increased BBB permeability, and is associated with rapid depletion of essential nutrients and oxygen (2-3). Only a few studies were designed in humans in order to compare the degree of BBB changes and the neurological outcome after a stroke. The most significant stage of BBB breakdown occurs in humans within 48-72 hours post infarction and is accompanied by increased brain edema volume.

The investigators performed a study on thirty patients with acute stroke of the middle cerebral artery using technetium-99m-DTPA brain SPECT (4). Tc-99m-DTPA (Diethylenetriamine- pentacetic acid) brain scintigraphy is a useful technique for the assessment of BBB disruption. Is has been used in the past to localize areas within the cranium which had been disrupted by infection, neoplasms, trauma or stroke. The study showed that the magnitude of disruption of the BBB was negatively correlated with the change in neurological status with a sensitivity of 95% and a specificity of 89%. Interestingly, a significant proportion of patients with stroke (23%) had no gross evidence of BBB disruption, all of them with very good prognosis.

It is unclear for how long the BBB remains disrupted after a stroke, and whether there is any correlation between the BBB permeability and recurrent ischemic events or delayed functional and neurological outcome after a stroke.

Aim of the study

In this study the investigators intend to explore the long term significance of BBB disruption on the clinical course and the rate of significant recurrent ischemic events in patients with a chronic stroke.

Patients and methods Inclusion criteria

Male and female patients at any age with a history of a large stroke in the territory of the middle cerebral artery, occurring 1-2 years ago or between 2-5 years ago.

Exlusion criteria

Methods:

40 patients will be recruited from the Neurological Outpatient Clinic of the Edith Wolfson Medical Center and from the Neurological Department.

For the SPECT study each patient will receive 740 MBq Tc-99m-DTPA and a SPECT study will be performed 60-90- minutes later. A dual head or a triple head gamma camera is usually used, equipped with high resolution collimators.

References

1. Persidsky Y, Ramirez SH, Haorah J, Kanmogne GD. Blood-brain barrier: structural components and function under physiologic and pathologic conditions. J Neuroimmune Pharmacol 2006;1:223-236.
2. del Zoppo GJ, Hallenbeck JM (2000) Advances in the vascular pathophysiology of ischemic stroke. Thromb Res 98:73-81
3. Petty MA, Wettstein JG (2001) Elements of cerebral microvascular ischaemia. Brain Res Rev 36:23-34
4. Lorberboym M, Lampl Y, Sadeh M. Correlation of 99mTc-DTPA SPECT of the blood-brain barrier with neurologic outcome after acute stroke. J Nucl Med 2003;44:1898-1904.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients at any age with a history of a large stroke in the territory of the middle cerebral artery, occurring 1-2 years ago or between 2-5 years ago.

Exclusion Criteria:

* Lacunar strokes,
* CNS lesions other than a stroke,
* unable to perform the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients at any age with a history of a large stroke in the territory of the middle cerebral artery, occurring 1-2 years ago or between 2-5 years ago.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2009-09; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Blood Brain Barrier permeability | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Wolfson Medical Center, Holon, Israel, Israel